CLINICAL TRIAL: NCT00472498
Title: Comparison on the Efficacy of a Monophasic, Manually Operated Defibrillator to That of a Biphasic Automatic External Defibrillator in the Hospital Setting.
Brief Title: Comparison on the Efficacy of a Monophasic
Acronym: AED
Status: Terminated | Type: Observational
Why Stopped: Terminated: No longer recruiting.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Samuel C. Dudley, Jr., Principal Investigator, Emory University
Other Study IDs: 206-2000
Record Dates: First submitted 2007-04-16; First posted 2007-05-11 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Biphasic Defibrillator
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Case:
  Patients resuscitated after 2001
- 2: Control:
  Patients who suffer cardiac arrests after 2001.

SUMMARY:
The central purpose of this study is to compare the clinical outcomes of patients who suffered a cardiac arrest while hospitalized at the VA and were resuscitated after biphasic defibrillators were implemented in 2001 to clinical outcomes of patients who suffered cardiac arrest before 2001.

DETAILED DESCRIPTION:
The central purpose of this study is to compare the clinical outcomes of patients who suffered a cardiac arrest while hospitalized at the VA and were resuscitated after biphasic defibrillators were implemented in 2001 to clinical outcomes of patients who suffered cardiac arrest before 2001.

This study will retrospectively collect and analyze clinical data related to the Atlanta VA Medical Center, a member of the National Registry of Cardiopulmonary Resuscitation, to assess clinical parameters in cardiac arrest survivors.

This study focuses on collecting data retrospectively in regard to cardiac arrest patients to discern what factors are playing a role in patient survival after cardiac arrest. Such data will help hospitals and physicians to improve quality of care in patients at risk for cardiac arrest as well as to implement strategies to reduce such events or improve management of these high-risk patients in order to save lives.

ELIGIBILITY:
Inclusion Criteria:

* Clinical outcomes of patients who suffered a cardiac arrest while hospitalized and were resuscitated after biphasic defibrillators were implemented in 2001 to clinical outcomes of patients who suffered cardiac arrest before 2001.

Exclusion Criteria:

Biphasic defibrillators were implemented Cardiac arrest before 2001

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized at the Atlanta VAMC hospital.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2005-06; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
s who suffered a cardiac arrest while hospitalized at the VA and were resuscitated | Information on patients who suffered cardiac arrest before 2001

SECONDARY OUTCOMES:
This study is observational. | Comparison before and after 2001

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C Dudley, MD, PhD, Principal Investigator — US Department of Veterans Affairs

REFERENCES:
- [Result] Zafari AM, Zarter SK, Heggen V, Wilson P, Taylor RA, Reddy K, Backscheider AG, Dudley SC Jr. A program encouraging early defibrillation results in improved in-hospital resuscitation efficacy. J Am Coll Cardiol. 2004 Aug 18;44(4):846-52. doi: 10.1016/j.jacc.2004.04.054. PMID 15312869
- [Result] Bloom HL, Shukrullah I, Cuellar JR, Lloyd MS, Dudley SC Jr, Zafari AM. Long-term survival after successful inhospital cardiac arrest resuscitation. Am Heart J. 2007 May;153(5):831-6. doi: 10.1016/j.ahj.2007.02.011. PMID 17452161